CLINICAL TRIAL: NCT00657982
Title: Phase II Study of RAD001 in a Neoadjuvant Setting in Men With Intermediate or High Risk Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr Raanan Berger, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-4616-RB-CTIL
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): RAD001 10 BID 6 weeks before definite treatment for localized prostate cancer
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — 10mg BID

SUMMARY:
The mechanisms responsible for the development of hormonal refractory prostate cancer (HRPC) have been elusive. Genetic inactivation/loss of the PTEN tumor suppressor gene occurs in 30-60% of advanced prostate cancers and in 20% of the localized form. Researchers hypothesize that PTEN loss is a landmark genetic event in prostate cancer progression into the fatal HRPC form. One consequence of PTEN loss is activation of the oncogenic Akt and phosphorylation of downstream Akt targets including mTOR. mTOR controls many important cellular processes including cell cycle regulation.

We propose to evaluate pharmacodynamic assessments of the mTOR inhibitor RAD001 in intermediate and high risk prostate cancer patients in the neoadjuvant setting. Patients will be admitted to 6 weeks treatment with RAD001 10 mg/day followed by either radical prostatectomy or radiotherapy combined with hormonal treatment. Immunohistochemistry with antibodies for phosphorylated p70S6K , pS6, Akt as well as antibodies for VEGF, BCL2 and PTEN in prostate cancer tissues before and after 6 weeks RAD001 treatment will be performed. Additionally, Patients will be evaluated by FDG-PET scan before (as baseline) and after RAD001 treatment. A link between mTOR signaling and glycolysis regulation was established and may provide a mechanism to assess drug-target interaction of RAD001 in prostate cancer.

The secondary endpoint of the trial will be to determine the response proportion to RAD001 treatment by assessing time to biochemical failure followed by radiation therapy or radical prostatectomy. The data will be compared to a matched cohort of high and intermediate-risk prostate cancer patients admitted to the same treatments modalities without receiving RAD001.

DETAILED DESCRIPTION:
Newly diagnosed patients with prostate cancer, with localized untreated disease must be at intermediate or high risk for disease relapse based on their PSA, Gleason score, and clinical stage. Before starting treatment, a baseline radiographic evaluation with FDG-PET and magnetic resonance imaging (MRI) will be performed. Biopsies will also be performed to obtain fresh tissue for molecular and gene expression assays. In patients with a positive FDG-PET scan at baseline, Treatment Day 1-14 will be with RAD001 10 mg/day alone. After performing post-RAD001 FDG-PET evaluation, treatment Day 15 will be equivalent of Treatment Day 1 of the trial in patients with negative FDG-PET scan at baseline.

In patients with a negative FDG-PET scan at baseline, Treatment Day 1 is the beginning of the Phase II trial of RAD001 combined with androgen ablation treatment.

Patients will be treated with RAD001 10 mg per day combined with androgen ablation therapy for 8 weeks depending on their ability to tolerate the drug. Radiographic and biologic assays will be repeated after 8 weeks, at which time patients will undergo prostatectomy or external beam radiation therapy (ERT). Second biopsy will be performed in patients admitted to ERT They will receive RAD001 up to the day of surgery or ERT to ascertain better tissue concentration of the drug. Gene expression profiling will also be evaluated at that time. The primary endpoint of this study is pharmacodynamic assessments of the effects of RAD001 in prostate cancer. However, the secondary endpoints of this study will define its true success. Specifically, the study will evaluate pharmacodynamic assessments of the effects of RAD001 in prostate cancer using novel applications of radiology, molecular biology, and genomics. These novel endpoints will be correlated with more established pathologic measures, such as microvessel density, apoptotic indexes, PTEN, phospho-AKT and phospho-p70S6K. MRI and 3-dimensional. PSA effects will also be assessed. Prostate cancer tissues from high risk prostate cancer patients admitted to neoadjuvant androgen ablation without RAD001 will serve as controls.

An ambitious aspect of this project is to examine gene expression alterations that occur in these patients. It will be technically challenging to get enough tissue by needle biopsies for gene array analysis. However, clearly, obtaining this information might be very useful in describing the full effects of RAD001 therapy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic documentation of adenocarcinoma of prostate Gleason grade 7-10
2. No evidence for lymph node or distant disease
3. No prior RT to pelvis or other regions
4. Age > 18 years
5. Performance status ECOG 0-1
6. ANC >1500/l
7. Hemoglobin > 9.0 g/dl
8. Platelets >100,000/l
9. Total Bilirubin <1.5 x upper limits of normal
10. AST or ALT < 3 x upper limits of normal
11. Creatinine < 1.5 x upper limits of normal
12. Electrolytes within 10% of normal Range
13. Cholesterol < 300

Exclusion Criteria:

1. Prior hormonal therapy
2. Prior RT to the pelvis
3. Currently active second malignancy other than non-melanoma skin cancer
4. Patients who have any severe and/or uncontrolled medical conditions such as

   1. Unstable angina pectoris, symptomatic congestive heart failure (New York heart association grade 2 or greater failure), myocardial infarction ≤ 6 months prior to randomization, serious uncontrolled cardiac arrhythmia
   2. Active or uncontrolled severe infection
   3. Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
   4. Severely impaired lung function
5. Evidence of bleeding diathesis or coagulopathy or need of administration of full-dose anti-coagulative(s)
6. Major surgical procedure, open biopsy or significant trauma within 28 days prior to day 1
7. Patients with active infection, including inflammation.
8. Prior therapy with mTOR inhibitors (sirolimus, temsirolimus, everolimus)
9. Uncontrolled diabetes mellitus as defined by fasting serum glucose >1.5
10. Patients receiving chronic treatment with corticosteroids or another immunosuppressive agent
11. Patients with a known history of HIV seropositivity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
PET-CT | 6 weeks

SECONDARY OUTCOMES:
PSA failure | 3-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Tel Hashomer, Israel